CLINICAL TRIAL: NCT06920745
Title: TRIClip CoverAge With Evidence Development (CED) Real-World Evidence (RWE) Study (TRICARE)
Brief Title: TriClip CED RWE Study
Acronym: TRICARE
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CL1028170
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Tricuspid Regurgitation
Keywords: TriClip; Coverage with Evidence Development; Tricuspid Transcatheter Edge-to-Edge Repair
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Treatment Group: Patients with symptomatic, severe or greater TR who received a T-TEER with the TriClip system
  Interventions: Device: The TriClip System
- Control Group: Patients with symptomatic, severe or greater TR without T-TEER

INTERVENTIONS:
Device: The TriClip System — The TriClip System
  Groups: Treatment Group

SUMMARY:
This Coverage with Evidence Development (CED) study evaluates the long-term health outcomes of patients with symptomatic, severe or greater Tricuspid Regurgitation who received a Tricuspid Transcatheter Edge-to-Edge Repair (T-TEER) procedure using the TriClip system.

DETAILED DESCRIPTION:
The TRICARE will assess 2-year effectiveness in patients with symptomatic, severe or greater TR who undergo Tricuspid Transcatheter Edge-to-Edge Repair (T-TEER) with the TriClip system, as compared to a contemporaneous control of patients without T-TEER.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age at time of implant
* Patients with symptomatic, severe or greater Tricuspid Regurgitation who have received the TriClip system (treatment group) or have not undergone T-TEER (control group)

Exclusion Criteria:

* Patients with less than severe Tricuspid Regurgitation
* Patients with a prior history of surgical or transcatheter tricuspid valve replacement
* Patients with a surgical or transcatheter aortic or mitral valve intervention within 90 days prior to index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world patients with symptomatic, severe or greater tricuspid regurgitation in the United States
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Composite of heart failure hospitalization or all-cause mortality | 2 years
  Compare the rate of composite endpoint at 2 years between the treatment and control groups.

SECONDARY OUTCOMES:
Tricuspid valve re-intervention | 2 years
  Report the rate at 2 years for the treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott, Santa Clara, California, United States